CLINICAL TRIAL: NCT06587932
Title: Effect of Brain Gym Exercises on Risk of Fall, Balance and Quality of Life in Obese Subjects
Brief Title: Brain Gym Exercises on Risk of Fall, Balance and Quality of Life in Obese Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Aya AbdElhady Ahmed Ali Elerian, EFFECT OF BRAIN GYM EXERCISES ON RISK OF FALL, BALANCE AND QUALITY OF LIFE IN OBESE SUBJECTS, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/005436
Record Dates: First submitted 2024-09-05; First posted 2024-09-19 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Obese Subjects

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (exprimental group) (Experimental): 16 subjects received brain gym exercises for 15-30 minutes per day, three times a week, for eight consecutive weeks . And traditional treatment in form of balance exercise included standing on one leg, standing in tandem mode, walking in a tandem mode (one foot in front of the other), walking on toes and heels, side walk, standing while one upper extremity and the opposite lower extremity were up, rotating the head from side to side, walking backwards for four steps, and shifting weight from one foot to the other. Periodic exercises were frequently performed for 45 min for 3 sessions per week for 8 weeks.
  Interventions: Other: brain gym exercises
- Group B (balance exercise): (Active Comparator): 16 subjects will receive traditional treatment in form of balance exercise included standing on one leg, standing in tandem mode, walking in a tandem mode (one foot in front of the other), walking on toes and heels, side walk, standing while one upper extremity and the opposite lower extremity were up, rotating the head from side to side, walking backwards for four steps, and shifting weight from one foot to the other. Periodic exercises were frequently performed for 45 min for 3 sessions per week for 8 weeks.
  Interventions: Other: Traditional treatments

INTERVENTIONS:
Other: brain gym exercises — It is comprised very easy body movements which have been designed to coax the two hemispheres of the brain.
  Arms: Group A (exprimental group)
Other: Traditional treatments — traditional treatment in form of balance training included standing on one leg, standing in tandem mode, walking in a tandem mode (one foot in front of the other), walking on toes and heels, side walk, standing while one upper extremity and the opposite lower extremity were up, rotating the head from side to side, walking backwards for four steps, and shifting weight from one foot to the other
  Arms: Group B (balance exercise):

SUMMARY:
This study will be done to answer the following question:

Do brain gym exercises have an effect on risk of fall, static balance, dynamic balance and risk of fall and quality of life in obese subjects?

DETAILED DESCRIPTION:
Obesity has now become a severe and inescapable worry for people of all generations. Obesity is associated with an excessive or inappropriate fat build-up that poses a health concern. A BMI of 25 or above is considered to be overweight, while a BMI of 30 is classified as obese. In 2017, nearly 4 million individuals died as a direct result of being overweight and obese, according to the global burden of sickness report. Postural equilibrium is required for us to function normally in our daily lives. The ability to manage the center of mass inside the base of support, which serves to maintain the body in balance, is characterized as equilibrium. Balance is described as the process of maintaining the body center of gravity within its support base, which necessitates regular modifications given by muscle activity and joint alignment . 1. Thirty-two obese subjects from both gender with age ranging from 18-50 years old . And BMI ≥ 30 kg/m2. They will be selected from faculty of physical therapy Kafr Elshikh university Group A (exprimental group): 16 subjects received brain gym exercises for 15-30 minutes per day, three times a week, for eight consecutive weeks . And traditional treatment in form of balance training included standing on one leg, standing in tandem mode, walking in a tandem mode (one foot in front of the other), walking on toes and heels, side walk, standing while one upper extremity and the opposite lower extremity were up, rotating the head from side to side, walking backwards for four steps, and shifting weight from one foot to the other. Periodic exercises were frequently performed for 45 min for 3 sessions per week for 8 weeks Group B (control group): 16 subjects will receive traditional treatment in form of balance training included standing on one leg, standing in tandem mode, walking in a tandem mode (one foot in front of the other), walking on toes and heels, side walk, standing while one upper extremity and the opposite lower extremity were up, rotating the head from side to side, walking backwards for four steps, and shifting weight from one foot to the other. Periodic exercises were frequently performed for 45 min for 3 sessions per week for 8 weeks

ELIGIBILITY:
Inclusion Criteria:1- Obese subjects from both gender age range from 18-50 years old (Cruz-Gomez et al., 2021) 2- BMI ≥ 30 kg/m2

-

Exclusion Criteria:neurological conditions affect the balance as:

* Alzheimer's disease
* Parkinson's disease
* Head injuries
* Peripheral neuropathy
* Headaches or migraines 2. lower limb injuries 3. Postural hypotension 4. Motion sickness 5. Diabetes mellitus 6. Pregnancy 7. Rheumatoid arthritis 8. osteoporosis

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
risk of fall | 6 months
  Modified Arabic version of Activities specific balance confidence scale to assess the risk of fall.
Static balance | 6 months
  Berg scale for static balance assessment
Dynamic balance | 6 months
  Balance check 636 device
Health related quality of life | 6 months
  Arabic version of WHO quality of life quationare bref to assess health related quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Maher A Elkeblawy, Phd, Study Chair — professor Cairo university; Yasser R Lasheen, Phd, Study Director — Assistant professor Cairo university
Locations (1):
- Cairo University, Cairo, Egypt